| Neuropathic Pain After Orchidectomy and Sex Reassignment Surgery (NPASRS) |
|---|
| ClinicalTrials.gov ID NCT 04538170 |
| Date of Initial Ethical Release: 23.10.2013 |
| Correspondence: |
| Barbara.Schlisio@med.uni-tuebingen.de |
| Department of Anaesthesiology and Intensive Care Medicine, Eberhard-Karls-University, Tuebingen, Germany |

### Background:

Phantom pain may occur after surgical removal of male reproductive organs. The indication for the surgery determines the physical and psychological predisposition of the patient that may differ between men who receive a tumor orchidectomy and those receiving gender reassignment surgery.

### Objective:

To determine whether patients experience phantom pain after gender reassignment surgery.

## Study protocol:

Transgender women who had undergone gender reassignment surgery in the Urology Clinic of the University of Tübingen and in the Surgical Clinic Munich-Bogenhausen should be retrospectively surveyed using written questionnaires. There should be at least 6 months between the survey and the surgical intervention for gender reassignment. Participation in the survey is pseudonymized and voluntary.

The control group includes men who had to undergo an orchiectomy for oncological indications. Here, too, there should be at least 6 months between the operation and the survey in order to record chronic pain and not postoperative pain.

### Study population:

The cohort size of the study is limited in that the gender reassignment surgery is a very rare procedure. We aim to include around 40 women in this group, with an estimated response rate of 80% for the questionnaires, so we want to write to at least 50 women. The control group (patients after oncological indicated orchiectomy) should include 145 men based on biometric considerations - with an estimated response rate of 60% in this group, we would write to 242 patients. For a difference of 20% considered relevant for the occurrence of phantom pain (approx. 25% share after oncological indicated orchidectomy, 5% after gender reassignment), a significance level of 5% with a power of 80% could be achieved.

Contact is made via the operating urological departments of the University Clinic Tübingen and the Surgical Clinic Munich-Bogenhausen. For this purpose, the patients are informed about the study (participant information). The questionnaire is pseudonymized and sent by post. Patients are asked to give their consent to the evaluation and publication of the research results in scientific journals. After receipt of the signed declaration of consent, the questionnaire will be scientifically evaluated.

Inclusion and exclusion criteria: Participation in this study is voluntary. You must be of legal age. The women and men should be able to give their consent and be able to fill out the form independently and without outside help.

# Test procedure:

Basic questionnaire to collect demographic data such as age, gender Pain detect questionnaire for the detection of neuropathic pain Record of phantom feelings and phantom pain through dichotomous questions Ability to cope with pain recorded by the FESV questionnaire Numerical rating scale (NRS) for recording the intensity of pain Health-related quality of life SF 12 Sexual satisfaction through dichotomous questions Incidence of surgical complications from dichotomous issues